CLINICAL TRIAL: NCT00593619
Title: A Randomized Double-Blind Safety Comparison of Intravenous Iron Dextran Versus Iron Sucrose in an Adult Non-Hemodialysis Outpatient Population: A Pilot Study
Brief Title: Trial Comparing the Safety of Two Different Intravenous Iron Formulations
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim Analysis and review by Data Safety Monitoring Board
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Ian H. Chin-Yee, Chair/Chief of Hematology, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSREB13767
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Iron Deficiency Anemia; Perioperative Blood Conservation
Keywords: Intravenous Iron; Safety; Perioperative; Iron deficiency; Non hemodialysis population; Perioperative blood conservation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — Iron-Dextran Complex; Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron Dextran (Active Comparator)
  Interventions: Drug: Iron dextran
- Iron Sucrose (Active Comparator)
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron dextran — 300mg in 250cc normal saline given over 2 hours
  Other Names: Infufer, Sandoz Canada Incorporated, DIN 02221780
  Arms: Iron Dextran
Drug: Iron sucrose — 300mg in 250cc normal saline given over 2 hours
  Other Names: Venofer, Luitpold Pharmaceuticals Inc., DIN 02243716
  Arms: Iron Sucrose

SUMMARY:
The purpose of this trial is to compare the safety profile using equal doses of intravenous iron dextran versus iron sucrose. The researchers hypothesize that significantly more patients receiving intravenous iron dextran (using the current intermediate molecular weight product) will have severe adverse outcomes than patients receiving iron sucrose in the adult non-hemodialysis outpatient population. Secondly, since these severe reactions may require additional nursing time and physician interventions that may negate any cost advantage of iron dextran, the researchers hypothesize that iron sucrose will be more cost-effective than iron dextran.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 100
* To be receiving intravenous iron

Exclusion Criteria:

* Age < 18
* Hemodialysis
* Previous exposure to intravenous iron
* Unable to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe adverse drug reactions (ADRs) | Immediate - during infusion

SECONDARY OUTCOMES:
Incidence of serious adverse drug reactions (ADRs) | Immediate and delayed - within 24hrs post infusion
Incidence of anaphylactic/anaphylactoid ADRs | Immediate - during infusion
Incidence of combined mild and moderate ADRs | Immediate - during infusion
Incidence of delayed ADRs | delayed - within 24hrs post infusion
Incidence of all-cause mortality | Immediate and delayed - within 24hrs post infusion
Physician and nursing time required to manage ADRs | Immediate and delayed - within 24hrs post infusion
Response in laboratory parameters | Within 1 month
Cost effectiveness | Completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Ian H Chin-Yee, MD, FRCPC, Principal Investigator — London Health Sciences Centre; Fiona E Ralley, MB ChB, FRCA, Principal Investigator — London Health Sciences Centre; Cyrus C Hsia, MD,FRCPC, Study Director — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada